CLINICAL TRIAL: NCT03579056
Title: Modeling of the Geriatric Multidisciplinary Meeting of the Angers University Hospital
Brief Title: GeRIatric Multidisciplinary Meeting
Acronym: GRIMM
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2017-06
Record Dates: First submitted 2017-10-26; First posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2017-10

CONDITIONS: Geriatric Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to develop a typology of patients referred to the Geriatric Multidisciplinary Meeting (GMM) according to their demographic and clinical profile.

The secondary objectives are:

* To distinguish the different types of answers given by the GMM according to the demands and situations.
* To study the factors associated with the orientation proposed by the GMM
* To examine the adequacy between the orientation proposed by the GMM and the pathway actually taken
* To compare the diagnoses made during the following year with the data collected during the GMM

DETAILED DESCRIPTION:
Increasing attention is paid to care pathways for elderly according to the principle of good care applied to the right patient at the right time and in the most appropriate care structure.

Since 2007, the geriatric mobile team (GMT) of the Angers University Hospital has formalized a geriatric multidisciplinary meeting (GMM) in connection with the geriatric network and branch of the geographical sector, in order to optimize the provision of care for elderly patients at the territorial level.

The weekly GMM brings together physicians from the geriatric department (GMT, acute care unit), memory center, long-term care and skilled nursing facilities, cognitive behavioral unit, psychiatry, retirement home, the local geriatric network of the city of Angers, the local information and coordination center, the home for autonomy and integration of Alzheimer patients (MAIA) and specialized Alzheimer (ESA) teams. Requests come either University Hospital services or from outside, via a standardized form. If necessary, additional data collection is carried out before the meeting by telephone with the patient, his family or the general practitioner. A letter explaining the decision of the GMM is sent to the applicant physician and to the general practitioner and recorded in the patient file.

Collegial guidance decisions within the health care system seem to follow implicit rules. Given the growing number of files presented, the investigators want to theorize the adopted mode of reflection.

ELIGIBILITY:
Inclusion Criteria:

* All the files discussed in GMM in the year 2015 following a request for geriatric care addressed to the Geriatrics department of the UH

Exclusion Criteria:

* No one

Min Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are recruited during the GMM of the University Hospital of Angers, France
Sampling Method: Non-Probability Sample
Enrollment: 734 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2017-09-04 (Actual)

PRIMARY OUTCOMES:
The demographic characteristics and medico-social data provided by the physician and the family at the time of the consultation request | baseline
  The demographic characteristics are age, sex, marital status, place of life, career, presence of un/formal assistance, …

SECONDARY OUTCOMES:
The answer given by the GMM | baseline
  This outcome is assessed by the guidance proposal issued by GMM
The orientation proposed by the GMM | baseline
  The recommendations made by GMM
The adequacy between the orientation proposed by the GMM and the pathway actually taken : back in the previous structure, hospitalization, reorientation, entry to a nursing home, other : | baseline and during the following year
  The course of care carried out at the Angers UH after the GMM
The diagnoses made during the following year with the data collected during the GMM : Alzheimer's disease, mixed dementia, body lewy, Parkinson's disease, frontotemporal dementia, vascular dementia, other | baseline and during the following year
  Diagnoses carried out at the Angers UH after the GMM

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University Hospital, Angers, France